CLINICAL TRIAL: NCT05954780
Title: A Non-interventional Study of Selinexor (Nexpovio®) in Combination With Bortezomib and Dexamethasone (SVd) in Patients With Relapsed or Refractory Multiple Myeloma (R/RMM)
Brief Title: Selinexor (Nexpovio®) (SVd) in Patients With Relapsed or Refractory Multiple Myeloma
Acronym: SEATTLE
Status: Active, not recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Menarini Stemline (Unknown); Climedo Health GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOM-090494
Record Dates: First submitted 2023-06-23; First posted 2023-07-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Selinexor; Bortezomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- second line and later lines therapy: Patients enrolled for second line or later lines therapy with selinexor in combination with bortezomib and dexamethasone.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Selinexor/bortezomib/dexamethasone according to Nexpovio® SmPC

SUMMARY:
The non-interventional study SEATTLE aims to answer open scientific questions regarding QoL and tolerability/safety and AE management of selinexor as well as effectiveness and dosing in clinical routine. Thus, SEATTLE will provide real-world evidence complementary to pivotal studies.

DETAILED DESCRIPTION:
Multiple myeloma (MM) accounts for approximately 10% of hematological malignancies. Since MM patients are elderly and often comorbid patients, risk-adapted treatment strategies to further improve outcome in is crucial.Selinexor, a potent, oral, SINE (selective inhibitors of nuclear exports) binds reversibly to XPO. This leads to nuclear localization and functional activation of tumor suppressor proteins, which further leads to suppression of nuclear factor κB activity, and reduction in oncoprotein mRNA translation. All this induces apoptosis of tumor cells. Since treatment options for MM are various and the most important factor is to keep or improve quality of life (QoL) of the patients, there is an urge for real-world clinical data of MM patients treated with selinexor in clinical routine. The objective of this non-interventional study is to evaluate QoL and tolerability/safety and AE management as well as effectiveness and dosing in adult patients with relapsed or refractory MM, which receive selinexor in combination with bortezomib and dexamethasone in the 2nd or later therapy line in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma
* Indication and decision for ≥2nd-line treatment with selinexor in combination with bortezomib and dexamethasone according to current selinexor SmPC as assessed by the treating physician
* Treatment decision before inclusion into this non-interventional study
* Willingness and ability to participate in the electronic patient-reported outcome (ePRO) module and answering of questionnaires
* Age ≥18 years
* Signed and dated informed consent form
* Inclusion before start of treatment (prospective inclusion)

Exclusion Criteria:

* Contraindications according to selinexor SmPC for patients with MM
* Participation in an interventional clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) with relapsed or refractory multiple myeloma and decision for treatment with selinexor in combination with bortezomib and dexamethasone (SVd) in ≥2nd therapy line
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of EORTC global health scale | Baseline, up to 40 months
  Change from baseline quality of life (QoL) over time for the global health scale of the EORTC QLQ- C30 questionnaire.

SECONDARY OUTCOMES:
Change from baseline of EORTC QLQ-C30 further scales | Baseline, up to 40 months
  Change from baseline in further scales of the EORTC QLQ-C30 questionnaire
Change from baseline of EORTC QLQ-MY20 further scales | Baseline, up to 30 days after selinexor treatment
  Change from baseline in further scales of the EORTC QLQ-MY20 questionnaire
Assessment of drug tolerability and safety | Baseline, up to 40 months
  Frequency of specific (serious) adverse drug reactions ((S)ADRs) (nausea, weight loss, diarrhea, vomiting, fatigue)
Adverse events (AEs) and serious adverse events (SAEs) according to NCI CTCAE | Baseline, up to 30 days after end of selinexor treatment
  Incidence of (serious) AEs ((S)AEs) as characterized by type, frequency, severity and seriousness.
Adverse drug reaction (ADR) and serious adverse drug reactions (SADR) | Baseline, up to 30 days after end of selinexor treatment
  Incidence of (serious) adverse drug reactions ((S)ADRs) as characterized by type, frequency, severity and seriousness.
Adverse events of special interest (AESI) | Baseline, up to 30 days after end of selinexor treatment
  Incidence of AEs of special interest defined as cataracts (new-onset cataracts and worsening of cataracts) and Acute cerebellar syndrome.
Changes in selinexor therapy | From date of selinexor treatment start, up to 40 months
  Frequency of treatment delays, no administrations (skips), discontinuation (withdrawn) of selinexor due to safety reasons
Effectiveness in routine treatment: Best response | Baseline, up to 40 months
  Frequencies of best response during selinexor therapy will be calculated using descriptive statistics.
Effectiveness in routine treatment: Overall response rate (ORR) | Baseline, up to 40 months
  ORR of patients will be calculated. ORR is defined as the proportion of patients achieving a complete response, very good partial response or partial response as best overall response. Patients without response measurement are considered non-responders.
Effectiveness in routine treatment: Disease control rate (DCR) | Baseline, up to 40 months
  DCR is defined as the proportion of patients achieving complete response, very good partial response, partial response, or stable disease as best response. Patients without response measurement are considered non-responders.
Effectiveness in routine treatment: Progression-free survival (PFS) | Baseline, up to 40 months
  PFS is defined as the time interval measured from the day of first selinexor administration to first progression or death, whichever comes first.
6 months PFS rate | Baseline, until 6 months after start of selinexor treatment
  PFS rates will be analysed 6 months after treatment start of selinexor
12 months PFS rate | Baseline, until 12 months after start of selinexor treatment
  PFS rates will be analysed 12 months after treatment start of selinexor
Effectiveness in routine treatment: Overall survival (OS) | Baseline, up to 40 months
  OS is defined as the time interval measured from the day of first selinexor administration to time of death from any cause.
6 months OS rate | Baseline, until 6 months after start of selinexor treatment
  OS rates will be analysed 6 and 12 months after treatment start of selinexor
12 months OS rate | Baseline, until 12 months after start of selinexor treatment
  OS rates will be analysed 6 and 12 months after treatment start of selinexor
Selinexor therapy: Dosing | Baseline, up to end of selinexor treatment
  Dose intensity during treatment (mg/m2 per week) will be analysed
Selinexor therapy: Frequency | Cycle 1, day 1
  Frequency of starting dose of selinexor (100 mg, 80 mg, 60 mg, other) will be analysed
Selinexor therapy: Dose reduction of starting dose | Cycle 1, day 1
  Reasons for reduced starting dose compared to SmPC will be analysed
Selinexor therapy: Dose changes | From date of second selinexor application, up to 40 months
  Reasons for dose reductions and dose re-escalation during treatment compared to previous dose
Previous therapies | Baseline
  Frequency of distinct previous therapies (systemic / radiation / transplantation)
Daratumumab-based previous therapies | Baseline
  Frequency of patients with daratumumab-based previous therapies
Treatment duration | From date of selinexor treatment start, up to 40 months
  Treatment duration of selinexor therapy
Subsequent antineoplastic therapies | From Date of end of selinexor treatment up to 40 months
  Frequency of distinct subsequent antineoplastic therapies.
Subsequent antineoplastic transplantations | From Date of end of selinexor treatment up to 40 months
  Frequency of distinct subsequent antineoplastic transplantations.
Subsequent antineoplastic radiations | From Date of end of selinexor treatment up to 40 months
  Frequency of distinct subsequent antineoplastic radiations.
Frequency of concomitant medication | Baseline up to 30 days after end of selinexor therapy
  Frequency of concomitant medication administered
Anti-emetic substances for AE treatment | Baseline up to 30 days after end of selinexor treatment
  Use of anti-emetic substances for AE treatment
Anti-emetic substances for prophylaxis | From date of selinexor treatment start, up to 40 months
  Use of anti-emetic substances for prophlaxis
Anti-diarrhea substances for AE treatment | Baseline up to 30 days after end of selinexor treatment
  Use of anti-diarrhea substances for AE treatment
Anti-diarrhea substances for prophylaxis | From date of selinexor treatment start, up to 40 months
  Use of anti-diarrhea substances for prophylaxis
Anti-emetic and anti-diarrhea substances for AE treatment | From date of selinexor treatment start, up to date of end of selinexor treatment
  Use of anti-emetic and anti-diarrhea substances for AE treatment
Anti-emetic and anti-diarrhea substances for prophylaxis | From date of selinexor treatment start, up to date of end of selinexor treatment
  Use of anti-emetic and anti-diarrhea substances for prophylaxis
Administration of Glucocorticoids and NK1 antagonist for prophylaxis | From date of selinexor treatment start, up to 40 months
  Frequency of glucocorticoids (i.e., dexamethasone given in addition to study medication) + NK1 antagonist administration used for prophylaxis.
Administration of NK1 + 5HT3 antagonist for prophylaxis | From date of selinexor treatment start, up to 40 months
  Frequency of NK1 + 5HT3 antagonist administration used for prophylaxis
Administration of Glucocorticoids and 5HT3 antagonist for prophylaxis | From date of selinexor treatment start, up to 40 months
  Frequency of glucocorticoids (i.e., dexamethasone given in addition to study medication) + 5HT3 antagonist administration used for prophylaxis.
Administration of Glucocorticoids, NK1 and 5HT3 antagonist for prophylaxis | From date of selinexor treatment start, up to 40 months
  Frequency of glucocorticoids (i.e., dexamethasone given in addition to study medication) + NK1 + 5HT3 antagonist administration used for prophylaxis.
Therapy decision | Baseline
  Assessment of parameters of therapy decision making.
Therapy choice | Baseline
  Frequency of distinct parameters affecting therapy choice.
Assessment of myeloma comorbidity index R-MCI | Baseline
  Assessment of R-MCI in all patients and patients with different starting doses
R-MCI risk groups | Baseline
  Frequency of R-MCI risk groups in all patients and according to different selinexor starting dosages (100 mg vs. 80 mg vs. 60 mg).

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Dechow, Prof. Dr., Study Chair — Gemeinschaftspraxis für Hämatologie und Onkologie GbR; Maria Krauth, Assoc. Prof. PD Dr., Study Chair — Universitätsklinikum AKH Wien
Locations (2):
- Medizinische Universität Wien, Universitätsklinik für Innere Medizin I, Vienna, Austria
- Gemeinschaftspraxis für Hämatologie und Onkologie GbR, Ravensburg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No